CLINICAL TRIAL: NCT05610748
Title: Implant-supported Rehabilitation of Atrophic Edentulous Sites With a Novel, Simplified Technique for Bone Augmentation or Soft Tissue Augmentation: a Randomized Trial
Brief Title: Implant-supported Rehabilitation With SPAL Technique or Soft Tissue Augmentation
Acronym: SPALvsSTA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Azienda USL Ferrara (Other Government)
Responsible Party: Principal Investigator, Leonardo Trombelli, Full Professor and Chair of Periodontology, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIN-RER_BU_2020_45
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Dehiscence; Alveolar Ridge Enlargement; Bone Loss, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: The study is designed as a single-blind, parallel-arm, randomized trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assignment of eligible patients to treatment will be recorded using sealed envelopes and will be disclosed to each clinical operator at the end of the screening appointment. The examiners will be kept blinded as to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-Periosteal Peri-implant Augmented Layer (SPAL) technique simultaneous to implant placement (Experimental): In patients assigned to the SPAL group, the management of the soft tissues will be performed according to the SPAL technique as originally described by Trombelli et al. (2018). Implant site preparation will be performed using a set of calibrated guided surgery steel burs under copious sterile saline irrigation. Implants will be placed, and a healing abutment will be positioned and screwed. The space underneath the periosteal layer will be then filled with a deproteinized bovine bone mineral (DBBM) graft. A sterile viscoelastic gel (SVG) based on polynucleotides and hyaluronic acid (REGENFAST®, Mastelli Srl, Sanremo, Italia) will be combined with the bone graft. The periosteal layer will be then secured to the oral flap by mean of 6/0 resorbable internal mattress sutures. SVG wil be placed underneath the mucosal layer and the latter will be coronally advanced and stabilized a using 6/0 resorbable internal mattress and sling sutures.
  Interventions: Procedure: Sub-Periosteal Peri-implant Augmented Layer technique
- Soft Tissue Augmentation (STA) simultaneous to implant placement (Active Comparator): In patients assigned to the STA group, flap management will be performed as described by Stefanini et al. (2016). Implant site preparation will be performed according to the same procedures described for the SPAL group. SVG will be placed underneath the buccal flap and the latter will be then released from tension by means of periosteal and muscular incisions, and will be coronally advanced and adapted to the healing abutment with a 6/0 resorbable sling suture. Interrupted sutures will be used to accomplish primary intention closure in the interproximal areas.
  Interventions: Procedure: Soft tissue augmentation

INTERVENTIONS:
Procedure: Sub-Periosteal Peri-implant Augmented Layer technique — In patients assigned to the SPAL group, the management of the soft tissues will be performed according to the SPAL technique as originally described by Trombelli et al. (2018). Implant site preparation will be performed using a set of calibrated guided surgery steel burs under copious sterile saline irrigation. Implants will be placed, and a healing abutment will be positioned and screwed. The space underneath the periosteal layer will be then filled with a deproteinized bovine bone mineral (DBBM) graft. A sterile viscoelastic gel (SVG) based on polynucleotides and hyaluronic acid (REGENFAST®, Mastelli Srl, Sanremo, Italia) will be combined with the bone graft. The periosteal layer will be then secured to the oral flap by mean of 6/0 resorbable internal mattress sutures. SVG wil be placed underneath the mucosal layer and the latter will be coronally advanced and stabilized a using 6/0 resorbable internal mattress and sling sutures.
  Other Names: SPAL
  Arms: Sub-Periosteal Peri-implant Augmented Layer (SPAL) technique simultaneous to implant placement
Procedure: Soft tissue augmentation — In patients assigned to the STA group, flap management will be performed as described by Stefanini et al. (2016). Implant site preparation will be performed according to the same procedures described for the SPAL group. SVG will be placed underneath the buccal flap and the latter will be then released from tension by means of periosteal and muscular incisions, and will be coronally advanced and adapted to the healing abutment with a 6/0 resorbable sling suture. Interrupted sutures will be used to accomplish primary intention closure in the interproximal areas.
  Other Names: STA
  Arms: Soft Tissue Augmentation (STA) simultaneous to implant placement

SUMMARY:
The primary aim of the present study is to compare the Sub-periosteal Peri-implant Augmented Layer (SPAL) technique and soft tissue augmentation (STA), performed simultaneously to implant placement, in terms of (i) implant survival rate and (ii) health/disease condition of the peri-implant tissues at 6 and 12 months following implant loading. The secondary aim of the project will be to compare the SPAL technique and STA in terms of intra- and post-operative morbidity.

The study is designed as a single-blind, parallel-arm, randomized clinical trial. Patients will be recruited and treated at the Operative Unit of Dentistry, Azienda Unità Sanitaria Locale (A.U.S.L.) of Ferrara, Italy, and one University center (Research Centre for the Study of Periodontal and Peri-implant Diseases, University of Ferrara, Italy). Each patient will contribute the study with one sextant ("experimental sextant"). Each eligible patient will be randomly assigned to receive SPAL technique or STA according to a computer-generated randomization list. Surgical procedures will be performed by experienced periodontal and implant surgeons. Two calibrated, blinded examiners will take care of the assessment of clinical and radiographic parameters, Case Report Form (CRF) filling, as well as data extraction from CRFs for the preparation of the study database.

The proportion of patients free from peri-implantitis at 12 months following loading will be the primary outcome variable of the study. The proportion of patients with complete resolution of the bone dehiscence (BD), dimensional variations and 12-months characteristics of BD, and patient-reported outcome measures will be the secondary outcomes. The design will test two hypotheses, with a non-inferiority trial in terms of primary outcome and a superiority trial in terms of secondary outcomes.

ELIGIBILITY:
Patient-specific inclusion criteria

* age≥21years;
* good physical status (ASA1 and ASA2 according to Physical Status Classification System) (American Society of Anesthesiologists, 2010);
* systemic and local conditions compatible with implant placement and experimental procedures;
* indication to a fixed, implant-supported prosthetic rehabilitation with hard or soft tissue reconstructive procedures as part of the comprehensive oral rehabilitation plan;
* patient willing and fully capable to comply with the study protocol.

Sextant-specific inclusion criteria

To be considered as experimental, a sextant will have to fulfill all the following criteria:

* including at least one healed (i.e., ≥ 6 months elapsed from tooth loss) edentulous site;
* horizontal dimension of the edentulous ridge compatible with the primary stability of an implant of at least 3.5 mm in diameter;
* expected peri-implant buccal BD characterized by a height (measured as the apico-coronal height of the exposed implant surface) ≤ 5 mm or a thin (< 1 mm) peri-implant buccal bone plate as diagnosed on tridimensional planning for guided implant placement.

Patient will not be eligible for the study if presenting at least one of the following exclusion criteria:

Patient-specific exclusion criteria

* current heavy smoking (≥20 cigarettes/day for ≥6 months prior to and at the time of the surgical procedure);
* untreated periodontal disease prior to implant placement;
* history of radiation therapy in the head and neck area;
* history of chemotherapy;
* systemic disease or conditions with a documented effect on bone metabolism and/or osseous healing;
* past (within 6 months prior to enrolment in the study) or current treatment with any medication with a documented effect on bone metabolism and/or osseous healing;
* documented allergy to dental materials involved in the experimental protocol;
* pregnancy or lactation;
* history of drug or alcohol abuse.

Moreover, participants immediately exited the study upon:

* request to withdraw from further participation;
* development of acute dental, peri-implant or oral conditions requiring treatment;
* development of conditions conflicting with the inclusion criteria listed above;
* failure to comply with study instructions/requirements.

Site specific exclusion criteria

* presence of either a buccal BD > 5 mm in depth or a thick (≥ 1 mm) peri-implant buccal bone plate as clinically assessed with a periodontal probe immediately after implant placement;
* presence of endodontic lesions at teeth adjacent to the implant site;
* previous bone augmentation/preservation procedures at the designated implant areas;
* need for vertical bone augmentation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients free from peri-implantitis | 12-month visit
  Proportion of patients free from peri-implantitis (diagnosed according to the criteria described by Berglundh et al. 2018) at 12 months following loading

SECONDARY OUTCOMES:
Complete resolution of bone dehiscence (BD) | 12-month visit
  Proportion of patients with complete resolution of BD as evaluated on CT/CBCT scan at 12 months following surgery
Changes in height and width of bone dehiscence (BD) | Pre-surgery and 12-month visits
  Variations in height and width of bone dehiscence (BD) (as evaluated on CT/CBCT scan) occurred between pre-surgery visit 12-month visits
Height and width of the residual bone dehiscence (BD) | 12-month visit
  Height and width of bone dehiscence (BD) as evaluated on CT/CBCT scan at 12-month visit
Pain | Day 0, +1, +2, +3, +4, +7 and +14 following surgery
  Level of pain recorded in the evening at day 0, +1, +2, +3, +4, +7 and +14 on a 100-mm visual analogue scale (VAS) ranging from "0-no pain" to "100-worst pain imaginable"
Dose of rescue anti-inflammatory drug | First 14 days following surgery
  Dosage of rescue anti-inflammatory drug (i.e. number of ibuprofen 600 mg tablets) and other types of medications taken from the day of surgery to the 14th postoperative day, as recorded daily on a medication diary.
Discomfort | Day 0, +1, +2, +3, +4, +7 and +14 following surgery
  Level of discomfort, as recorded at day 0 (evening), +1, +2, +3, +4, +7 and +14 on a 5-point rating scale ranging from "no discomfort" to "very high discomfort"
Limitations in daily functions | Day 0, +1, +2, +3, +4, +7 and +14 following surgery
  Limitations in daily functions (i.e., swallowing, continuing daily activities, eating, speaking, opening the mouth, sleeping), as recorded at day 0 (evening), +1, +2, +3, +4, +7 and +14 on a 5-point rating scale ranging from "no limitations" to "unable to eat a lot of types of food" (for the "eating" item), and from "not at all difficult" to "extremely difficult" (for the other items)
Incidence of postoperative signs and symptoms | Day 0, +1, +2, +3, +4, +7 and +14 following surgery
  Incidence of postoperative signs and symptoms (i.e., swelling, nausea, bruising, bad taste/smell) at day 0 (evening), +1, +2, +3, +4, +7 and +14
Willingness to undergo the same type of surgery | Day +14 following surgery
  Willingness to undergo the same type of surgery, recorded at day +14 on a 4-point rating scale ranging from "no problem to repeat surgery if needed" to "I will never undergo this type of surgery again."

CONTACTS AND LOCATIONS:
Locations (1):
- Polo Odontoiatrico, Ferrara, Italy